CLINICAL TRIAL: NCT06946329
Title: Mechanistic and Functional Outcomes of WATERinMOTION Aquatic Therapy in Obese Men With Knee Osteoarthritis: A Randomized Controlled Trial With 6-Month Follow-Up
Brief Title: WATERinMOTION Aquatic Therapy in Obese Men With Knee Osteoarthritis
Acronym: WATERinMOTION
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sistan and Baluchestan (Other)
Responsible Party: Principal Investigator, Mohammadreza Rezaeipour, Assoc.Prof.Dr., University of Sistan and Baluchestan
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 9378-1403
Record Dates: First submitted 2025-04-19; First posted 2025-04-27 (Actual); Last update posted 2025-04-27 (Actual); Status verified 2025-04

CONDITIONS: Osteoarthritis; Knee; Obesity
Keywords: Aquatic Therapy; Exercise Therapy; Quality of Life; Biomarkers; Wearable Electronic Devices
MeSH Terms: conditions — Osteoarthritis; Obesity | interventions — Aquatic Therapy

STUDY DESIGN:
Intervention Model Description: Parallel Assignment
Who Masked: Outcomes Assessor
Masking Description: Single-blind (outcome assessors only; participants/instructors unblinded due to intervention nature).
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Aquatic Exercise (Experimental): Supervised WATERinMOTION sessions (60 mins, 3x/week) in heated pool. Focus on progressive resistance and mobility exercises.
  Interventions: Behavioral: Aquatic Exercise
- Land-Based Rehabilitation (Active Comparator): Matched frequency/duration land-based program emphasizing core stabilization and low-impact aerobics.
  Interventions: Behavioral: Land-Based Rehabilitation

INTERVENTIONS:
Behavioral: Aquatic Exercise — Supervised WATERinMOTION sessions (60 mins, 3x/week) in heated pool. Focus on progressive resistance and mobility exercises.
  Arms: Aquatic Exercise
Behavioral: Land-Based Rehabilitation — Matched frequency/duration land-based program emphasizing core stabilization and low-impact aerobics.
  Arms: Land-Based Rehabilitation

SUMMARY:
This RCT evaluates whether WATERinMOTION aquatic therapy improves pain, function, and quality of life more effectively than land-based exercise in obese men with knee osteoarthritis (OA). We will assess clinical outcomes (WOMAC), serum biomarkers (COMP, IL-6), and real-world activity (accelerometry) at baseline, 8 weeks, and 6 months.

DETAILED DESCRIPTION:
100 participants (BMI ≥30, age 45-65, radiographic knee OA) will be randomized to:

Aquatic group: 24 sessions over 8 weeks (3x/week) in 32°C water, progressing from buoyancy-assisted to resistance exercises.

Land group: Matched duration/intensity land-based rehabilitation. Primary outcomes: WOMAC pain/function. Secondary outcomes: SF-36 quality of life, serum COMP, 6-minute walk test, and accelerometer-measured step count.

ELIGIBILITY:
Inclusion Criteria:

* Males aged 45-65
* BMI ≥30 kg/m²
* Radiographic knee OA (Kellgren-Lawrence grade 2-3)
* WOMAC pain score ≥25/50

Exclusion Criteria:

* Inflammatory arthritis (e.g., rheumatoid)
* Intra-articular injections within 3 months
* Contraindications to aquatic exercise

Ages: 45 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Males aged 45-65
Enrollment: 100 (Estimated)
Dates: Start 2024-03-01 (Actual); Primary Completion 2024-09-30 (Actual); Study Completion 2025-05-01 (Estimated)

PRIMARY OUTCOMES:
WOMAC Pain Subscale | Baseline, 8 weeks, 6 months
  Change from baseline in WOMAC pain score (0-20 scale).
WOMAC Function Subscale | Baseline, 8 weeks, 6 months
  Change in functional disability (0-68 scale).

SECONDARY OUTCOMES:
SF-36 Quality of Life | Baseline, 8 weeks, 6 months
  Physical/Mental Component Summaries (0-100).
Serum COMP | Baseline, 8 weeks
  Change in cartilage oligomeric matrix protein (ng/mL).
Daily Step Count | Continuous over 8 weeks
  Measured via ActiGraph GT9X accelerometer.

CONTACTS AND LOCATIONS:
Overall Officials: Mohammadreza Rezaeipour, MD,PhD, Study Director — Assoc.Prof.Dr. of University of Sistan and Baluchestan, Zahedan, Iran
Locations (1):
- Sport Sciences Department, Zahedan, Sistan and Baluchestan, Iran

IPD SHARING:
Plan to Share IPD: No
Privacy concerns (sensitive health data of overweight/obese men). Lack of pre-specified data-sharing plan in ethics approval.